CLINICAL TRIAL: NCT05470751
Title: A Multi-centre Prospective Observational Study of the User Experience of Catheterisation and Quality of Life in Patients Prescribed GentleCath™ for Men Intermittent Catheter With FeelClean™ Technology
Brief Title: GentleCath™ for Men Intermittent Catheter With FeelClean™ Technology
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-21-425
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Bladder Outlet Obstruction; Multiple Sclerosis; Cauda Equina Syndrome; Enlarged Prostate With Lower Urinary Tract Symptoms; Parkinson Disease; Lower Urinary Tract Symptoms; Detrusor Underactivity; Spinal Cord Injuries
Keywords: neurogenic bladder; intermittent self-catherterisation; pain; bladder outflow obstruction
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Multiple Sclerosis; Cauda Equina Syndrome; Parkinson Disease; Lower Urinary Tract Symptoms; Urinary Bladder, Underactive; Spinal Cord Injuries; Urinary Bladder, Neurogenic; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Intermittent self-catheterisation — Self-catheterising with GC Male and Glide Male with Feelclean technology

SUMMARY:
Male self catherterisng observational study.

DETAILED DESCRIPTION:
This is a multicentre, prospective international observational study. Male patients in the UK, USA and France performing self-catheterisation will be asked to participate in this study. The subjects will be asked to use the GentleCath™ Intermittent Catheter with FeelClean™ Technology as per their normal routine. They will be asked to record when and where they catheterise. At the baseline, during and on completion of the study, the subjects will be asked to complete Difficulty in Catheterisation plus Intermittent Catheter related Quality of Life Questionnaires.

Difficulty during catheterisation and quality of life will be assessed using the ICDQ and ISC-Q validated questionnaires during catheterisation at the start of the study before use of GentleCath™ Air has commenced (D0) and on day 1 (D1), day 15 (D15), day 30 (D30), day 45 (D45) and day 60 (D60) transcribed in a collecting record provided for this purpose. Compliance and catheter use will also be assessed.

Patient confidence regarding reduced stickiness plus related risk of urethral injury and resultant bleeding or infection will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* • Adult male (aged 18 years and over)

  * Diagnosed with a neurological lower urinary tract dysfunction due to either spinal cord injury, Multiple Sclerosis, Parkinson's Syndrome, Cauda equina syndrome Or Diagnosed with bladder outflow obstruction secondary to benign prostate enlargement Or Diagnosed with detrusor underactivity
  * Performing single use clean intermittent self-catheterisation (ISC) at least twice a day
  * Willing to undergo training with GC Trainer video prior to use of catheter
  * Provided fully informed consent and has sufficient understanding of English or French
  * Sufficient dexterity to use GentleCath™ Air for Men intermittent including ability to open packaging
  * Intact urethral sensation of catheterisation
  * Willing to use only the GentleCath™ Air intermittent catheter for the full duration of the study (60-days)
  * Subject has a valid email address so the Investigator can send links to study questionnaires and the subject has access to a web enabled device

Exclusion Criteria:

* • Participation in another related urological study

  * Unable to perform ISC unaided
  * Already prescribed the GentleCath™ Air Intermittent Catheter
  * Absent urethral or perineal sensation
  * Unwilling to undergo training with GC Trainer prior to use of catheter
  * Insufficient dexterity to use GentleCath™ Air Intermittent Catheter and or packaging
  * Suffering from a symptomatic UTI (Urinary Tract Infections) at the time of inclusion or in the preceding 6-weeks
  * Undergoing surgical treatment during the period of the study
  * Performing catheterisation for urethral stricture

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be able to insert catheter into a penile urethra
Study Population: Adult males who self-catheterise
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
To assess difficulty during catheterisation and quality of life using the ICDQ and ISC-Q validated questionnaires during catheterisation | 60 days
  To assess difficulty during catheterisation and quality of life using the ICDQ and ISC-Q

SECONDARY OUTCOMES:
To assess patient confidence regarding reduced stickiness plus related risk of urethral injury and resultant bleeding or infection | 60 days
  To assess patient confidence regarding reduced stickiness plus related risk of urethral
To assess compliance with the self-catheterization for the study duration | 60 days
  To assess compliance with the self-catheterization for the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Chris Harding, Principal Investigator — Site Investigator - Newcastle
Locations (16):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - Trustees of The University of Pennsylvania | Penn Urology Washington Square, Philadelphia, Pennsylvania
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux | Pellegrin Hospital - Urology Department, Bordeaux
  - Assistance Publique Hopitaux de Paris | Pitie Salpetriere University Hospital - Urology Department, Paris
- United Kingdom (12):
  - Stockport NHS Foundation Trust | Stepping Hill Hospital - Research and Innovation Department, Stockport, Cheshire
  - Broomfield Hospital, Chelmsford, Essex
  - Mid and South Essex NHS Foundation Trust | Southend University Hospital - Research & Development, Southend-on-Sea, Essex
  - Aneurin Bevan University Health Board | Royal Gwent Hospital - Clinical Research Centre, Newport, Gwent
  - Southampton General Hospital, Southampton, Hampshire
  - Kent and Canterbury Hospital | Renal Research Delivery Team, Canterbury, Kent
  - Newcastle upon Tyne Hospitals NHS Foundation Trust | Freeman Hospital - Urology Department, Newcastle, Newcastle Upon Tyne
  - Sunderland Royal Hospital, Sunderland, Tyne & Wear
  - North Bristol NHS Trust | Southmead Hospital - Research and Development - Urology Department, Bristol, Westbury-on-Trym
  - Mid Yorkshire Teaching NHS Trust | Pinderfields Hospital - Yorkshire Regional Spinal Injuries Centre, Wakefield, Yorkshire
  - Guy's and St Thomas' Foundation Trust | Guy's Hospital - Transplant, Renal and Urology Research, London
  - King's College Hospital NHS Foundation Trust | King's College Hospital - Renal Research Department, London

IPD SHARING:
Plan to Share IPD: No